CLINICAL TRIAL: NCT05608616
Title: COVID-19 and Pregnancy Maternal and Fetal Outcomes,A Retrospective Cross Sectional Study
Brief Title: Maternal and Fetal Outcomes in Pregnant Women With COVID -19,a Cross Sectional Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mostafa Mohammed Refaay El shemy, Lecturer at Obstetrics and Gynecology department, Cairo University
Other Study IDs: COVID-19 and pregnancy
Record Dates: First submitted 2022-11-05; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The spread of a new coronavirus (SARS-CoV-2) from Wuhan, China, has been fast, and the World Health Organization (WHO) declared a pandemic on March 11th, 2020 .It has now spread worldwide and is one of the most severe public health threats.The clinical characteristics of COVID-19 and the likelihood of transmission vertically or during delivery in pregnant women are still unknown.

DETAILED DESCRIPTION:
In this cross sectional study,the following questions require immediate attention: whether COVID-19 symptoms in pregnant women differ from symptoms in non-pregnant women; whether disease complications and mortality rates are higher in pregnant women than in non-pregnant women; and whether there is a risk of premature delivery, foetal mortality, or even vertical transmission of the disease. These questions must be answered in order to plan optimal obstetrical management for pregnant women with COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women of any gestational age with confirmed COVID 19 diagnosis attended and admitted at inpatient ward for management and follow up from April 2020 to December 2021at Kasr El Ainy hospital,Cairo university

Exclusion Criteria:

* there is no exclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A retrospective analysis of prospectively collected data of pregnant women confirmed as COVID-19 infected.
  Maternal and fetal morbidities and adverse obstetrical outcomes among those with COVID-19 will be analyzed.
  Maternal outcomes will include:Venous thromboembolic events,pregnancy outcome,mode of delivery,frequency of admission to ICU,need for assistive ventilation,mortality rate Fetal outcomes will include:Frequency of NICU admission,Preterm birth,Intrauterine growth restriction,Intrauterine fetal death,Congenital fetal malformations.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Outcomes of Pregnancy with COVID-19 | 32 months
  Prevalence of maternal and fetal morbidities and adverse obstetrical outcomes among pregnant women with COVID-19 diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt